CLINICAL TRIAL: NCT06823089
Title: Early Feasibility Study of Cartilage Defect Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cytex Therapeutics, Inc. (Other)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-0001
Record Dates: First submitted 2025-01-22; First posted 2025-02-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Hip; Femoroacetabular Impingement; Osteonecrosis; Trauma Related Injuries; Avascular Necrosis of Bone of Hip; Avascular Necrosis of Bone
Keywords: articular cartilage; hip; impingement; osteochondral; resurfacing; hip resurfacing; hip replacement; osteonecrosis; avascular necrosis
MeSH Terms: conditions — Osteoarthritis, Hip; Femoracetabular Impingement; Osteonecrosis

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, non-comparative, single-arm, open-label, multicenter, clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Investigational Arm (Experimental): The investigation device for this study will be the ReNew Hip Implant.
  Interventions: Device: ReNew Hip Implant

INTERVENTIONS:
Device: ReNew Hip Implant — Surgical Intervention

SUMMARY:
Any patient aged 14 or older up to 64 years of age with hip disease, resulting in loss of articular cartilage integrity on the femoral head (e.g., femoroacetabular impingement or other structural deformity), has failed conservative care, and is a candidate for surgical intervention to treat.

DETAILED DESCRIPTION:
When patients suffer from arthritis in the hip joint and fail conservative treatment, the standard surgical approach is total joint arthroplasty, where the joint is entirely removed and replaced with artificial materials. While this procedure is suitable for less active or older individuals, it is not ideal for younger, more active patients. Despite this, the number of total hip replacements in younger patients is increasing, requiring significant lifestyle adjustments to extend the implant's lifespan. Even with these efforts, most patients will face at least one total joint revision in their lifetime, each carrying an increased risk of complications and decreased patient satisfaction. As a result, total hip replacements are generally not recommended for patients aged 40 to 65 who experience activity-limiting symptoms and have exhausted conservative treatments.

The Cytex device offers an alternative treatment option for this patient population - those suffering from hip osteoarthritis (OA), unresponsive to conservative care, yet considered too young or active for total joint replacement. Notably, the Cytex implant preserves all pre-existing healthy bone stock, unlike traditional total hip resurfacing or arthroplasty procedures, allowing for future revision to conventional resurfacing or arthroplasty if needed.

The investigational device for this study, the ReNew Hip Implant, is a bioabsorbable, highly porous implant designed with mechanical properties that closely mimic those of healthy articular cartilage. The implant features a bicomponent structure, combining a biomimetic 3D woven textile with a porous 3D-printed framework.

ELIGIBILITY:
Inclusion Criteria:

1. At least 14 years of age to no older than 64 years of age Subjects 14-21 years of age must have radiographic evidence of epiphyseal closure in the hip joint
2. BMI < 35
3. Failed at least 6 weeks of conservative treatment (e.g., anti-inflammatory pain medications, physical therapy, injections)
4. Duration of symptoms consistent with intra-articular disease (i.e., groin, lateral and/or posterior hip pain) that have persisted for at least 3 months)
5. Loss of articular cartilage integrity (~1 - 6 cm^2 in area) on the femoral head (confirmed by MRI), without an opposing lesion, that can be treated with a single ReNew Hip Implant
6. Radiographic assessment with joint space width > 2 mm (verified by x-ray)
7. Meets an acceptable preoperative medical clearance and is free of conditions that would pose excessive operative risk, in the opinion of the investigator
8. Given consent to participate in the study
9. Able to understand the purpose of the study, his/her role, and is available for follow-up for the duration of the study:

   1. Subject has signed an IRB (Institutional Review Board) approved Informed Consent Form agreeing to participate in the extension study after the nature, scope, and possible consequences of the study have been explained in an understandable form
   2. Subject is able to fully understand the purpose of the study, his/her role as a participant in the study, and plans to be available through five years post-operative follow-up

Exclusion Criteria:

1. Current users of nicotine in any form (e.g., cigarettes, e- cigarettes/vaping, chewing tobacco, nicotine patches, gum, lozenges), or individuals who have discontinued nicotine use less than 30 days prior to screening.
2. Type 1 or Type 2 Diabetes
3. Systemic steroid use in the 3 months prior to screening
4. Coxa plana, coxa magna, or proximal femoral focal deficiency on the femoral head that would result in implant mismatch of the femoral head contour
5. Any acute or chronic condition that would limit the ability of the patient to participate in the study (e.g., COPD, congestive heart failure),
6. Bleeding disorders
7. Current cancer (with the exception of non-melanoma skin cancer)
8. Pregnancy or planning to become pregnant during the study period
9. Active infection or sepsis
10. History of local hip infection
11. Known metastatic or neoplastic disease
12. Conditions that may interfere with implant survival or outcomes (e.g., severe dysplasia)
13. Life expectancy less than 2 years
14. Intra-articular therapy within 3 months of enrollment
15. Inadequate bone stock (as determined by SCORE or MORES assessment) to support the device
16. Femoral head is:

    1. outside of the 46 - 56 mm range in either anteroposterior diameter or lateral diameters or
    2. an aspherical head deformity that results in contour mismatch of 16a
17. Moderate to severe renal insufficiency
18. Emotional or neurological condition that would preempt ability or willingness to participate in the study
19. Above the knee amputation of the contralateral or ipsilateral leg
20. Known allergies to the components of the device (polycaprolactone)
21. Is a prisoner

Ages: 14 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
To establish initial safety (adverse events and device related serious adverse events) and effectiveness (pain and function) of the ReNew Hip Implant | 6, 12, and 60 months
  Incidence rate of all adverse events including general adverse events, procedure related events and device related events.
  Incidence rate of device-related serious adverse events
The international Hip Outcome Tool-33 (iHOT-33) | 6, 12, and 60 months
  Difference demonstrated between pre-op and post-op iHOT-33

SECONDARY OUTCOMES:
Radiographic | 6, 12, and 60 months
  Imaging MRI of operative joint assessing the implant by MOCART 2.0 (modified), implant placement, joint effusion, and osteophytosis
Kaplan Meier survivorship | 12, 24, and 60 months post-surgery
  Kaplan Meier survivorship of the ReNew Hip Implant in terms of revision and / or radiological migration
Patient Reported Outcome Measures | 6, 12, 24, and 60 months post-surgery
  Difference demonstrated between pre-op and the post-op of all PROMs (mHHS, UCLA, PROMIS)
Health economic outcomes | Time Frame: Intra-operative
  Surgical blood loss; Measured in ml blood
Health economic outcomes | Time Frame: Hospital admission to discharge
  Length of hospital stay; Measure of days spent in hospital
Health economic outcomes | Intra-operative
  Operative time - first incision into skin to time when last suture is applied
Health economic outcomes | Time Frame: Up to 60 months
  Re-hospitalizations for hip issues; Re-hospitalizations number of re-admissions to hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- [Background] Roemer FW, Hunter DJ, Winterstein A, Li L, Kim YJ, Cibere J, Mamisch TC, Guermazi A. Hip Osteoarthritis MRI Scoring System (HOAMS): reliability and associations with radiographic and clinical findings. Osteoarthritis Cartilage. 2011 Aug;19(8):946-62. doi: 10.1016/j.joca.2011.04.003. Epub 2011 Apr 20. PMID 21550411
- [Background] Gold SL, Burge AJ, Potter HG. MRI of hip cartilage: joint morphology, structure, and composition. Clin Orthop Relat Res. 2012 Dec;470(12):3321-31. doi: 10.1007/s11999-012-2403-7. PMID 22723242